CLINICAL TRIAL: NCT00158431
Title: Arthroscopic Surgery Versus Non-surgical Treatment of Osteoarthritis of the Knee
Brief Title: Surgery Versus no Surgery for OA of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sharon Griffin, Research Coordinator, Fowler Kennedy Sport Medicine Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FKSMC-CIHR-1; CIHR MCT-15227 (Other Grant/Funding Number: Canadian Instititute for Health Research)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; randomized trial; knee; quality of life
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroscopy; Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopy plus Medical Management (Active Comparator): Arthroscopic Surgery of the Knee plus the optimized medical management including physiotherapy, education, medication, etc
  Interventions: Procedure: Arthroscopy plus Medical Management; Other: Medical Management
- Medical Management (No Intervention): Optimized Medical management including physiotherapy, education, medication, etc

INTERVENTIONS:
Procedure: Arthroscopy plus Medical Management — Arthroscopic Surgery
  Arms: Arthroscopy plus Medical Management
Other: Medical Management — education, optimized medication, weight loss where needed, HA or cortisone injections if needed, physiotherapy
  Arms: Arthroscopy plus Medical Management

SUMMARY:
The purpose of this trial is to evaluate the effectiveness of arthroscopy (lavage and debridement) in conjunction with the best available non-surgical treatment versus the best available non-surgical treatment alone (medication, health education and physical therapy) in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Osteoarthritis is estimated to affect half of the adult population, and by the age of 75 years, it is anticipated that 85 of 100 elderly patients will have some form of this disease. Osteoarthritis (OA) is characterized by moderate to severe pain that limits functional ability. It is suspected that the causes of this debilitating pain include irritation of the synovium, excessive subchondral bone forces and raised intra-arterial pressure. The knee is the most commonly affected weight-bearing joint. Osteoarthritis has a great social impact, as the second most common reason for work disability in the United States. The prevalence of OA is expected to increase in the coming years due to increased longevity, increased proportion of the population over the age of 75 years, and increased diagnostic ability.

Rather than further evaluations of different forms of arthroscopic surgery (ie lavage vs debridement vs abrasion) in the treatment of knee OA, we feel it is important to establish the efficacy of this technology compared to the best non-surgical treatment alone.

This is an evaluator- blinded, phase III, single-centre, group sequential randomized controlled trial in patients with osteoarthritis of the knee.

Treatment effectiveness is based upon patients' disease specific quality of life at 2 years using the Western Ontario McMaster (WOMAC) Osteoarthritis Index. In addition patients' physical function and cost effectiveness are being assessed. Costs will be estimated from the perspectives of the health care system, the patient,family, and society and will include the use of hospital and other resources as well as the economic implications of lost workdays associated with these alternative treatments.

This randomized clinical trial will provide high quality evidence to determine what the role of this expensive treatment is in the overall management of OA.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic or secondary osteoarthritis of the knee as diagnosed by Altman et al 2 classification tree -83 percent sensitivity, 93percent specificity
2. Grades 2 to 4 severity of OA by radiographic evaluation- modified Kellgren and Lawrence grading system
3. Age greater than 18.

Exclusion Criteria:

1. Inflammatory or post-infection arthritis of the knee
2. Previous arthroscopy for treatment of knee OA
3. Isolated medial compartment OA Grade 3-4 with greater than 5 degrees mechanical varus -ideal candidate for high tibial osteotomy
4. Isolated lateral compartment OA Grade III-IV with greater than 5 degrees mechanical valgus -ideal candidate for high tibial osteotomy or distal femoral osteotomy
5. Grade 4 OA in at least 2 compartments and over 60 years of age -ideal candidate for total knee arthroplasty
6. Cortico-steroid injection within the last three months.
7. Major neurological deficit
8. Major medical illness -life expectancy less than 2 years or with unacceptably high operative risk.
9. Pregnant
10. Unable to speak or read English
11. Psychiatric illness that limits informed consent
12. Unwilling to be followed for 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 1999-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To compare between the two treatment groups the patients' disease-specific quality of life at 2 years using the Western Ontario McMaster (WOMAC) osteoarthritis index and | 2 years

SECONDARY OUTCOMES:
SF-36,Mactar, Arthritis Self-Efficacy Scale, Standard Gamble Utility Measure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Fowler, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada

REFERENCES:
- [Background] Altman RD, Fries JF, Bloch DA, Carstens J, Cooke TD, Genant H, Gofton P, Groth H, McShane DJ, Murphy WA, et al. Radiographic assessment of progression in osteoarthritis. Arthritis Rheum. 1987 Nov;30(11):1214-25. doi: 10.1002/art.1780301103. PMID 3689459
- [Background] Baumgaertner MR, Cannon WD Jr, Vittori JM, Schmidt ES, Maurer RC. Arthroscopic debridement of the arthritic knee. Clin Orthop Relat Res. 1990 Apr;(253):197-202. PMID 2317974
- [Background] Bert JM. Role of abrasion arthroplasty and debridement in the management of osteoarthritis of the knee. Rheum Dis Clin North Am. 1993 Aug;19(3):725-39. PMID 8210584
- [Background] Blackburn WD Jr, Bernreuter WK, Rominger M, Loose LL. Arthroscopic evaluation of knee articular cartilage: a comparison with plain radiographs and magnetic resonance imaging. J Rheumatol. 1994 Apr;21(4):675-9. PMID 8035392
- [Background] Brandt KD. Should osteoarthritis be treated with nonsteroidal anti-inflammatory drugs? Rheum Dis Clin North Am. 1993 Aug;19(3):697-712. PMID 8210582
- [Background] Brandt KD, Fife RS, Braunstein EM, Katz B. Radiographic grading of the severity of knee osteoarthritis: relation of the Kellgren and Lawrence grade to a grade based on joint space narrowing, and correlation with arthroscopic evidence of articular cartilage degeneration. Arthritis Rheum. 1991 Nov;34(11):1381-6. doi: 10.1002/art.1780341106. PMID 1953815
- [Background] Brief AA, Maurer SG, Di Cesare PE. Use of glucosamine and chondroitin sulfate in the management of osteoarthritis. J Am Acad Orthop Surg. 2001 Mar-Apr;9(2):71-8. doi: 10.5435/00124635-200103000-00001. PMID 11281631
- [Background] Burks RT. Arthroscopy and degenerative arthritis of the knee: a review of the literature. Arthroscopy. 1990;6(1):43-7. doi: 10.1016/0749-8063(90)90096-v. No abstract available. PMID 2178619
- [Background] Chandler EJ. Abrasion arthroplasty of the knee. Contemporary Orthopaedics; 1121-1985
- [Background] Chang RW, Falconer J, Stulberg SD, Arnold WJ, Manheim LM, Dyer AR. A randomized, controlled trial of arthroscopic surgery versus closed-needle joint lavage for patients with osteoarthritis of the knee. Arthritis Rheum. 1993 Mar;36(3):289-96. doi: 10.1002/art.1780360302. PMID 8452573
- [Background] Deyle GD, Henderson NE, Matekel RL, Ryder MG, Garber MB, Allison SC. Effectiveness of manual physical therapy and exercise in osteoarthritis of the knee. A randomized, controlled trial. Ann Intern Med. 2000 Feb 1;132(3):173-81. doi: 10.7326/0003-4819-132-3-200002010-00002. PMID 10651597
- [Background] Dieppe P, Cushnaghan J, Jasani MK, McCrae F, Watt I. A two-year, placebo-controlled trial of non-steroidal anti-inflammatory therapy in osteoarthritis of the knee joint. Br J Rheumatol. 1993 Jul;32(7):595-600. doi: 10.1093/rheumatology/32.7.595. PMID 8339132
- [Background] Edelson R, Burks RT, Bloebaum RD. Short-term effects of knee washout for osteoarthritis. Am J Sports Med. 1995 May-Jun;23(3):345-9. doi: 10.1177/036354659502300317. PMID 7661265
- [Background] Felson DT, Zhang Y, Anthony JM, Naimark A, Anderson JJ. Weight loss reduces the risk for symptomatic knee osteoarthritis in women. The Framingham Study. Ann Intern Med. 1992 Apr 1;116(7):535-9. doi: 10.7326/0003-4819-116-7-535. PMID 1543306
- [Background] Fife RS, Brandt KD, Braunstein EM, Katz BP, Shelbourne KD, Kalasinski LA, Ryan S. Relationship between arthroscopic evidence of cartilage damage and radiographic evidence of joint space narrowing in early osteoarthritis of the knee. Arthritis Rheum. 1991 Apr;34(4):377-82. doi: 10.1002/art.1780340402. PMID 2012624
- [Background] Fisher NM, Gresham GE, Abrams M, Hicks J, Horrigan D, Pendergast DR. Quantitative effects of physical therapy on muscular and functional performance in subjects with osteoarthritis of the knees. Arch Phys Med Rehabil. 1993 Aug;74(8):840-7. doi: 10.1016/0003-9993(93)90011-x. PMID 8347069
- [Background] Fisher NM, Pendergast DR, Gresham GE, Calkins E. Muscle rehabilitation: its effect on muscular and functional performance of patients with knee osteoarthritis. Arch Phys Med Rehabil. 1991 May;72(6):367-74. PMID 2059102
- [Background] Goldman RT, Scuderi GR, Kelly MA. Arthroscopic treatment of the degenerative knee in older athletes. Clin Sports Med. 1997 Jan;16(1):51-68. doi: 10.1016/s0278-5919(05)70007-7. PMID 9012561
- [Background] Graf J, Neusel E, Schneider E, Niethard FU. Intra-articular treatment with hyaluronic acid in osteoarthritis of the knee joint: a controlled clinical trial versus mucopolysaccharide polysulfuric acid ester. Clin Exp Rheumatol. 1993 Jul-Aug;11(4):367-72. PMID 8403580
- [Background] Harwin SF. Arthroscopic debridement for osteoarthritis of the knee: predictors of patient satisfaction. Arthroscopy. 1999 Mar;15(2):142-6. doi: 10.1053/ar.1999.v15.015014. PMID 10210070
- [Background] Jones AC, Doherty M. The treatment of osteoarthritis. Br J Clin Pharmacol. 1992 Apr;33(4):357-63. doi: 10.1111/j.1365-2125.1992.tb04052.x. PMID 1576063
- [Background] Ike RW, Arnold WJ, Rothschild EW, Shaw HL. Tidal irrigation versus conservative medical management in patients with osteoarthritis of the knee: a prospective randomized study. Tidal Irrigation Cooperating Group. J Rheumatol. 1992 May;19(5):772-9. PMID 1613709
- [Background] Kim HK, Moran ME, Salter RB. The potential for regeneration of articular cartilage in defects created by chondral shaving and subchondral abrasion. An experimental investigation in rabbits. J Bone Joint Surg Am. 1991 Oct;73(9):1301-15. PMID 1918112
- [Background] Kirkley A, Webster-Bogaert S, Litchfield R, Amendola A, MacDonald S, McCalden R, Fowler P. The effect of bracing on varus gonarthrosis. J Bone Joint Surg Am. 1999 Apr;81(4):539-48. doi: 10.2106/00004623-199904000-00012. PMID 10225800
- [Background] Kovar PA, Allegrante JP, MacKenzie CR, Peterson MG, Gutin B, Charlson ME. Supervised fitness walking in patients with osteoarthritis of the knee. A randomized, controlled trial. Ann Intern Med. 1992 Apr 1;116(7):529-34. doi: 10.7326/0003-4819-116-7-529. PMID 1543305
- [Background] Kramer JS, Yelin EH, Epstein WV. Social and economic impacts of four musculoskeletal conditions. A study using national community-based data. Arthritis Rheum. 1983 Jul;26(7):901-7. doi: 10.1002/art.1780260712. PMID 6223644
- [Background] Leardini G, Mattara L, Franceschini M, Perbellini A. Intra-articular treatment of knee osteoarthritis. A comparative study between hyaluronic acid and 6-methyl prednisolone acetate. Clin Exp Rheumatol. 1991 Jul-Aug;9(4):375-81. PMID 1934686
- [Background] Lequesne M, Brandt K, Bellamy N, Moskowitz R, Menkes CJ, Pelletier JP, Altman R. Guidelines for testing slow acting drugs in osteoarthritis. J Rheumatol Suppl. 1994 Sep;41:65-71; discussion 72-3. PMID 7799389
- [Background] Liachenko, A. Cox-2 inhibitors offer hope to arthritis sufferers. Geriatrics and Aging 2(3):13, 1999.
- [Background] Livesley PJ, Doherty M, Needoff M, Moulton A. Arthroscopic lavage of osteoarthritic knees. J Bone Joint Surg Br. 1991 Nov;73(6):922-6. doi: 10.1302/0301-620X.73B6.1720118.
- [Background] Manek NJ, Lane NE. Osteoarthritis: current concepts in diagnosis and management. Am Fam Physician. 2000 Mar 15;61(6):1795-804. PMID 10750883
- [Background] Matheson AJ, Perry CM. Glucosamine: a review of its use in the management of osteoarthritis. Drugs Aging. 2003;20(14):1041-60. doi: 10.2165/00002512-200320140-00004. PMID 14651444
- [Background] McGinty JB, Johnson LL, Jackson RW, McBryde AM, Goodfellow JW. Uses and abuses of arthroscopy: a symposium. J Bone Joint Surg Am. 1992 Dec;74(10):1563-77. No abstract available. PMID 1469020
- [Background] McLaren AC, Blokker CP, Fowler PJ, Roth JN, Rock MG. Arthroscopic debridement of the knee for osteoarthrosis. Can J Surg. 1991 Dec;34(6):595-8. PMID 1747839
- [Background] Merchan EC, Galindo E. Arthroscope-guided surgery versus nonoperative treatment for limited degenerative osteoarthritis of the femorotibial joint in patients over 50 years of age: a prospective comparative study. Arthroscopy. 1993;9(6):663-7. doi: 10.1016/s0749-8063(05)80503-1. PMID 8305102
- [Background] Minor MA, Hewett JE, Webel RR, Anderson SK, Kay DR. Efficacy of physical conditioning exercise in patients with rheumatoid arthritis and osteoarthritis. Arthritis Rheum. 1989 Nov;32(11):1396-405. doi: 10.1002/anr.1780321108. PMID 2818656
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735
- [Background] Novak PJ, Bach BR Jr. Selection criteria for knee arthroscopy in the osteoarthritic patient. Orthop Rev. 1993 Jul;22(7):798-804. PMID 8414655
- [Background] Rand JA. Arthroscopic management of degenerative meniscus tears in patients with degenerative arthritis. Arthroscopy. 1985;1(4):253-8. doi: 10.1016/s0749-8063(85)80093-1. PMID 3841640
- [Background] Rashad S, Revell P, Hemingway A, Low F, Rainsford K, Walker F. Effect of non-steroidal anti-inflammatory drugs on the course of osteoarthritis. Lancet. 1989 Sep 2;2(8662):519-22. doi: 10.1016/s0140-6736(89)90651-x. PMID 2570233
- [Background] Reginster JY, Deroisy R, Rovati LC, Lee RL, Lejeune E, Bruyere O, Giacovelli G, Henrotin Y, Dacre JE, Gossett C. Long-term effects of glucosamine sulphate on osteoarthritis progression: a randomised, placebo-controlled clinical trial. Lancet. 2001 Jan 27;357(9252):251-6. doi: 10.1016/S0140-6736(00)03610-2. PMID 11214126
- [Background] Ruane R, Griffiths P. Glucosamine therapy compared to ibuprofen for joint pain. Br J Community Nurs. 2002 Mar;7(3):148-52. doi: 10.12968/bjcn.2002.7.3.10214. PMID 11904551
- [Background] Salisbury RB, Nottage WM, Gardner V. The effect of alignment on results in arthroscopic debridement of the degenerative knee. Clin Orthop Relat Res. 1985 Sep;(198):268-72. PMID 4028560
- [Background] Sprague NF 3rd. Arthroscopic debridement for degenerative knee joint disease. Clin Orthop Relat Res. 1981 Oct;(160):118-23. PMID 7285411
- [Background] Timoney JM, Kneisl JS, Barrack RL, Alexander AH. Arthroscopy update #6. Arthroscopy in the osteoarthritic knee. Long-term follow-up. Orthop Rev. 1990 Apr;19(4):371-3, 376-9. PMID 2185456
- [Background] van Baar ME, Assendelft WJ, Dekker J, Oostendorp RA, Bijlsma JW. Effectiveness of exercise therapy in patients with osteoarthritis of the hip or knee: a systematic review of randomized clinical trials. Arthritis Rheum. 1999 Jul;42(7):1361-9. doi: 10.1002/1529-0131(199907)42:73.0.CO;2-9. PMID 10403263
- [Background] van Tienen TG, Heijkants RG, de Groot JH, Pennings AJ, Poole AR, Veth RP, Buma P. Presence and mechanism of knee articular cartilage degeneration after meniscal reconstruction in dogs. Osteoarthritis Cartilage. 2003 Jan;11(1):78-84. doi: 10.1053/joca.2002.0870. PMID 12505490
- [Background] Vaughn BK, Eberle RW, and Rayburn SM. Outcome of arthroscopically-aided debridement of the knee as an alternative to total knee arthroplasty. 1997.
- [Background] Yang SS, Nisonson B. Arthroscopic surgery of the knee in the geriatric patient. Clin Orthop Relat Res. 1995 Jul;(316):50-8. PMID 7634724
- [Background] Myllyla V, Finkelstein H, Mayer L. Arthroscopy of the knee joint. Journal of Bone and Joint Surgery; 16255-1934
- [Background] Richards RN, Lonergan RP. Arthroscopic surgery for relief of pain in the osteoarthritic knee. Orthopedics. 1984 Nov;7(11):1705-7. doi: 10.3928/0147-7447-19841101-08. PMID 24822615
- [Derived] Birmingham TB, Primeau CA, Shariff SZ, Reid JNS, Marsh JD, Lam M, Dixon SN, Giffin JR, Willits KR, Litchfield RB, Feagan BG, Fowler PJ. Incidence of Total Knee Arthroplasty After Arthroscopic Surgery for Knee Osteoarthritis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e246578. doi: 10.1001/jamanetworkopen.2024.6578. PMID 38635272
- [Derived] Marsh JD, Birmingham TB, Giffin JR, Isaranuwatchai W, Hoch JS, Feagan BG, Litchfield R, Willits K, Fowler P. Cost-effectiveness analysis of arthroscopic surgery compared with non-operative management for osteoarthritis of the knee. BMJ Open. 2016 Jan 12;6(1):e009949. doi: 10.1136/bmjopen-2015-009949. PMID 26758265
- [Derived] Kirkley A, Birmingham TB, Litchfield RB, Giffin JR, Willits KR, Wong CJ, Feagan BG, Donner A, Griffin SH, D'Ascanio LM, Pope JE, Fowler PJ. A randomized trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2008 Sep 11;359(11):1097-107. doi: 10.1056/NEJMoa0708333. PMID 18784099